CLINICAL TRIAL: NCT04601038
Title: Phase II Trial of CORT108297 to Attenuate the Effects of Acute Stress in the Allocortex (CORT-X)
Brief Title: Trial of CORT108297 to Attenuate the Effects of Acute Stress in the Allocortex (CORT-X)
Acronym: CORT-X
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Private Philanthropic Funds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00227116
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Memory Impairment
Keywords: Stress; Memory loss; Dementia; Alzheimer's disease; Cognitive; Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Memory Disorders; Dementia | interventions — CORT 108297

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MCI (Other): Individuals with mild cognitive impairment due to Alzheimer's disease
  Interventions: Drug: CORT108297; Drug: Placebo
- Cognitively Normal (Other): Individuals who are cognitively normal but who are at risk for Alzheimer's disease
  Interventions: Drug: CORT108297; Drug: Placebo

INTERVENTIONS:
Drug: CORT108297 — 120mg of a selective glucocorticoid receptor antagonist, taken as 2 tablets daily for 2 weeks
Drug: Placebo — Placebo taken as 2 tablets daily for 2 weeks

SUMMARY:
CORT-X will examine if mitigation of stress-mediated pathogenesis of Alzheimer's disease (AD) is a feasible target for intervention in individuals at risk for this disease. This single-site (Baltimore, Maryland) phase II clinical trial is a 2-week, randomized, placebo-controlled crossover study of the effects of the selective glucocorticoid receptor antagonist, CORT108297, on cognitive test performance in 26 individuals with mild cognitive impairment (MCI) due to AD and in 26 cognitively normal individuals with an increased risk for AD due to family history, genetics, and/or subjective memory complaints. All subjects will participate in a brief stressor (public speaking and mental arithmetic) and provide saliva samples so investigators can measure stress hormone response. Then, following 2 weeks of treatment with placebo or CORT108297, in counterbalanced order, participants will complete cognitive tests assessing memory and executive function. All study participants will receive CORT108297 and placebo over the course of this 10-week trial that requires 6 in-person study visits. The primary aims will compare the effects of CORT108297 to placebo on cognitive test performance in individuals with MCI due to AD and in individuals at risk for AD, and describe the side effects of CORT108297 in study participants. Secondary aims will identify subject characteristics that predict positive response to study drug.

ELIGIBILITY:
Individuals must meet criteria for mild cognitive impairment due to Alzheimer's disease according to National Institute on Aging (NIA)/Alzheimer's Association recommendations OR be cognitively normal based on clinical and cognitive assessment in the Enrollment Visit and have at least one of the following risk factors for AD:

* Known to have at least 1 apolipoprotein E (APOE) ε4 allele;
* Subjective cognitive concerns with a T score < 40 on the Multifactorial Memory Questionnaire Satisfaction Scale;
* A first-degree relative with dementia.

Inclusion Criteria for all subjects:

* At least 55 years of age;
* Body mass index >17 and <30;
* Post-menopausal (if female)
* Non-smoker;
* Availability of a study partner who has frequent contact with the subject (10+ hours/week in person and by telephone), and is able to provide an independent evaluation of functioning;
* Native English speaker;
* Good general health with no disease expected to interfere with the study;
* Willing and able to participate for the duration of the study.

Exclusion Criteria for all subjects:

* Participation in a therapeutic clinical trial at any time during the study;
* Abnormal corrected QT interval using Bazett's formula (QTcB; defined as > 450 ms for men and > 470 ms for women) as determined on ECG;
* Any significant neurologic disease other than suspected incipient Alzheimer's disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities, including lacunes in critical memory structures including the hippocampus and parahippocampal cortex;
* Major depression, bipolar disorder within the past 1 year;
* History of alcohol or drug dependence;
* Any significant systemic illness or unstable medical condition, which could lead to difficulty complying with the protocol;
* General surgery within the last 3 months;
* Sensory impairment (poor vision or hearing) significant enough to interfere with ability to provide valid cognitive test data;
* Treatment within the last six months with antidepressants, neuroleptics, sedative hypnotics, or glucocorticoids;
* Treatment within the last six months with medications metabolized by the CYP2C9 or CYP2C19 enzymes, most notably clopidogrel and proton pump inhibitors;
* Concurrent use of a CYP3A inhibitor, including grapefruit juice, and St. John's Wort;
* Exceptions to these guidelines may be considered on a case-by-case basis at the discretion of the PI.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Memory as assessed by pattern separation task performance after 2 weeks of treatment with CORT108297 | After 2 weeks of treatment
  Percent of correct responses to the "lure" items on the pattern separation task, with 100% indicating a perfect score
Memory as assessed by the Hopkins Verbal Learning Test-Revised Edition (HVLT-R) after 2 weeks of treatment with CORT108297 | After 2 weeks of treatment
  Total number of words recalled in trials 1, 2, 3, and the delayed recall trial of the HVLT-R, with scores ranging from 0 (no words recalled) to 48 (all 12 words recalled after each of the trials)
Executive functioning as assessed by the Trail Making Test (TMT), part B after 2 weeks of treatment with CORT108297 | After 2 weeks of treatment
  Number of seconds required to complete part B of the TMT, with lower scores indicating better performance
Executive functioning as assessed by the Digit Span Task (digit span backwards) after 2 weeks of treatment with CORT108297 | After 2 weeks of treatment
  Total number of correct responses on the backwards trials of the Digit Span Task, with scores ranging from 0 (no trials correct) to 14 (perfect score)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Munro, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States